CLINICAL TRIAL: NCT00622921
Title: Couples-based Behavioral Psychotherapy for Male Patients With Posttraumatic Stress Disorder and Alcohol Dependence
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0711003228; 0711003228
Record Dates: First submitted 2008-02-13; First posted 2008-02-25 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: PTSD; Alcohol Dependence
Keywords: PTSD; alcohol dependence
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Couples-based behavioral psychotherapy
  Interventions: Behavioral: Couples-based behavioral psychotherapy

INTERVENTIONS:
Behavioral: Couples-based behavioral psychotherapy — 12 weeks of Couples-based behavioral psychotherapy

SUMMARY:
Purpose: Phase I focus groups with clinicians and patients will gather qualitative data to focus and inform the content of Phase II. In Phase II, 12 weeks of psychotherapy will be offered to evaluate feasibility and potential efficacy of a couples-based, integrated treatment for men with PTSD and alcohol dependence.

Hypotheses: We predict that this experimental psychotherapy, Partners Encouraging Abstinence and Coping with Emotions (PEACE), will reduce patient drinking, reduce PTSD symptoms, and improve relationship functioning.

ELIGIBILITY:
Inclusion Criteria:

* Male patients
* One to six weeks of abstinence from alcohol and other drugs
* Both partners agree to stated goals of abstinence from alcohol and drugs, reduction of PTSD symptoms, and relationship improvement
* Current diagnoses of both alcohol dependence and PTSD
* Receiving treatment for one or both disorders
* Functionally able to participate in outpatient treatment as determined by P.I. "Functionally able" includes access to transportation.
* Alcohol is "drug of choice" (History of other drugs acceptable)
* Married or cohabiting in stable relationship for at least 6 months. Separated couples may participate if attempting to reconcile
* Patient willing to sign release of information allowing researchers to communicate with patient's clinician regarding treatment goals

Exclusion Criteria:

* Spouse or partner also has an alcohol or drug problem as determined by P.I. based on report by patient or partner or as revealed on Alcohol Use Disorders Identification Test (AUDIT) or the Drug Abuse Screening Test (DAST) given to partner at intake assessment
* Mental retardation or learning disorder by clinician report or patient chart
* Psychotic disorder as determined by patient's chart or SCID
* Patient currently receiving methadone or another opiate agonist by patient report or chart
* Current fear of partner or history of severe domestic violence in the past year. An example of severe violence would be a couple reporting an episode of violence that required medical attention. Such couples will be excluded from the study and referred to domestic violence treatment. Couples who have experienced mild to moderate domestic violence may participate in Phase II of the study.

Ages: 21 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-02; Primary Completion 2012-02 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
PTSD symptoms, Alcohol use | 12 weeks

SECONDARY OUTCOMES:
relationship functioning | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ismene L Petrakis, MD, Principal Investigator — Yale University
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States